CLINICAL TRIAL: NCT06041061
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial Evaluating the Efficacy, Safety, and Immunogenicity of a 14- Valent Recombinant Human Papillomavirus Vaccine (SCT1000) in Healthy Women Aged 18-45 Years
Brief Title: A Study to Evaluate the Efficacy, Safety, and Immunogenicity of SCT1000 in Healthy Women Aged 18-45 Years
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government); Henan Center for Disease Control and Prevention (Other Government); Sichuan Center for Disease Control and Prevention (Other Government); Centers for Disease Control and Prevention, China (Other Government); Yunnan Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCT1000-03
Record Dates: First submitted 2023-08-13; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: HPV InfectioN; HPV-Related Carcinoma
Keywords: HPV; Vaccine
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Recombinant 14-Valent Human Papillomavirus Vaccine (Types 6,11,16,18,31,33,35,39, 45,51,52,56,58,59) （Insect Cell）
Who Masked: Participant, Investigator
Masking Description: Blinds for randomized subjects and drug coding blinds will be generated and stored by an independent third party. Immunogenic subgroup blind maintenance: The subgroup information shall not be disclosed to the testing personnel. The serological test results report of the immunogenic subgroup shall be received by non-blind personnel independent of the project team, and the personnel designated by the data management unit shall be responsible for checking the blind data. Before the study is unblinded, the serum results should not be disclosed to the relevant personnel to ensure the blindness of serological test results.
  In order to ensure the implementation of the blind method, iDMC will be established in this experiment. At the time of the interim analysis, iDMC was responsible for completing the primary efficacy markers and safety assessment, while the sponsors, investigators, and project staff of the trial remained blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the experiment vaccine
  Interventions: Biological: Recombinant 14-Valent Human Papillomavirus Vaccine（Insect Cell）
- placebo (Placebo Comparator): According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Recombinant 14-Valent Human Papillomavirus Vaccine（Insect Cell） — According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the experiment vaccine
  Arms: experiment group
Biological: placebo — According to the 0, 2, and 6 months immunization program, intramuscular injection of the upper arm deltoid muscle, 3 doses of the placebo
  Arms: placebo

SUMMARY:
A total of 18000 healthy women aged 18-45 years old were divided into three age groups: 18-26 years old, 27-35 years old, and 36-45 years old. The experimental group and the placebo group were randomly assigned in a ratio of 1:1. All subjects enrolled in the upper arm deltoid muscle were injected with 3 doses of test vaccine or placebo according to the 0, 2, and 6 months immunization program.

DETAILED DESCRIPTION:
Introduction: SCT1000 is a recombinant 14-valent human papillomavirus vaccine (insect cell) that covers all 12 WHO-recognized high-risk oncogenic HPV subtypes Indications are for the prevention of cervical, vulvar, vaginal, and anal cancers, and genital warts caused by HPV6, HPV11 and HPV11 in females 9-45 years of age, as well as intraepithelial neoplasia and AIS. Intraepithelial neoplasia and AIS and genital warts due to HPV6 and HPV11.

Aim:To evaluate the protective efficacy of 3 doses of HPV vaccine (SCT1000) for the prevention of HPV type 6,11,16,18,31,33,35,39,45,51,52,56,58,59-associated lesions in healthy females aged 18-45 years compared with placebo.

Design: A Multicenter, Randomized, Double-blind, Placebo-controlled phase III Clinical trial Subject Information: a total of 18000 healthy women aged 18-45 years selected by inclusion and exclusion criteria.

Cluster situation: a ratio of 1:1 between the experimental group and the placebo group.

End point index: relative index with efficacy, safety, and immunogenicity of SCT1000

ELIGIBILITY:
Inclusion Criteria:

* 1. Females who are at least 18 years old and less than 46 years old (i.e., 18 to 45 years old).

  2. Subjects sign a written informed consent form (ICF) to participate in the trial voluntarily, and are able to fully understand the trial procedures, the risks of participating in the trial, and the alternative interventions available to them if they do not participate in the trial.

  3. Be able to read, understand and complete the diary/contact card. 4. Be in good health as judged by the history interview and physical examination.

  5. Have a history of sexual behavior prior to enrollment. 6.*Avoid sexual intercourse (including same-sex or opposite-sex anal, vaginal, or genital/genital contact) and avoid vaginal douching, vaginal cleansing, or the use of vaginal medications or preparations for 48 hours prior to any visit that includes sample collection.

  7. Subjects who are not breastfeeding at the time of enrollment and who have used effective contraception from the time of their last menstrual period until enrollment in the study, and who understand and agree to use effective contraception from the first day of enrollment until 1 month after the last vaccination.

  8.* Those with axillary body temperature <37.3°C on the day of enrollment. 9. Note: Subjects who do not meet the *enrollment criteria are allowed to be screened again, but the enrollment criteria still need to be confirmed again at the time of enrollment.

Exclusion Criteria:

* 1. *Positive urine pregnancy test or pregnancy (including ectopic pregnancy) that has ended less than 6 weeks ago.

  2. Prior vaccination with a marketed HPV vaccine or already enrolled in a clinical trial of another HPV vaccine or have plans to receive a non-study HPV vaccine during the study period.

  3. Have a prior history of cervical cancer screening abnormalities or lesions [including HPV DNA positivity, squamous intraepithelial lesions (SIL) or atypical squamous cells of undetermined significance (ASC-US), atypical squamous epithelial cells-without the exception of high grade squamous intraepithelial lesions (ASC-H), atypical glandular cells (AGC), or have cervical intraepithelial neoplasia (CIN), adenocarcinoma in situ (AIS) or cervical cancer]. ) or cervical cancer, etc.].

  4. Previous or current anal or genital disease (e.g. vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts, vulvar, vaginal, and anal cancers) 5. Previous total hysterectomy or pelvic radiation therapy or severe developmental abnormalities of the cervix/vagina.

  6. History of drug or alcohol abuse or dependence in the last year. 7. Have hypertension or diabetes mellitus that cannot be controlled and stabilized with pharmacological interventions.

  8. Subjects with a history of severe allergic reactions to any vaccine or medication requiring medical intervention (e.g., anaphylaxis, anaphylactic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, localized anaphylactic necrotic reaction [Arthus reaction], etc.).

  9. Currently immunocompromised or diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, tuberculosis, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune disease.

  10. Previous splenectomy or impaired splenic function. 11. Currently receiving or have received the following immunosuppressive therapies in the last year: radiation therapy, cyclophosphamide, imidazathioprine, methotrexate, as well as chemotherapy, cyclosporine, leflunomide, tumor necrosis factor-alpha antagonists, monoclonal antibody therapies, intravenous gammaglobulin, anti-lymphocytic serums, or other therapies that are known to interfere with immunity 12. Current treatment with systemic corticosteroids or 2 or more courses of high-dose glucocorticoids lasting one week in the year prior to enrollment. The use of nasal inhaled glucocorticoids or topical short-term topical application on the skin may not be excluded.

  13. Receipt of any immunoglobulin product or blood product within 3 months prior to vaccination, or planning to receive such similar products during the study period from Day 1 to Month 7.

  14. * Inactivated/recombinant/nucleic acid vaccine, etc. (non-attenuated) within 14 days prior to vaccination or live attenuated vaccine within 28 days prior to vaccination.

  15. Contraindication to intramuscular injection such as thrombocytopenia or other coagulation disorders.

  16. *Blood donation within 1 week prior to vaccination or planning to donate blood between Day 1 and Month 7 of study participation.

  17. Participation in other experimental clinical studies or studies with unregistered products (drugs or vaccines) or collection of cervical specimens within 3 months prior to vaccination.

  18. Inability to follow trial procedures or planned relocation during the study.

  19. *Fever (axillary temperature ≥37.3°C) within 3 days prior to vaccination or any acute illness requiring systemic antibiotic or antiviral therapy within the past 5 days.

  20. *Clinical signs/symptoms suggestive of acute reproductive tract infection (e.g. acute vulvovaginitis/vaginitis/cervicitis [including purulent cervicitis], etc.) during gynecological examination.

  21. * Being in the menstrual period (sampling should be done 2 days after the end of menstruation).

  22. Have an active neurological/psychiatric/psychological disorder that prevents compliance with the study requirements.

  23. Have other abnormalities, conditions that may confound the results of the study, or conditions that are not in the best interest of the subject and may be excluded as determined by the investigator.

  24. Note: Subjects who meet *exclusion criteria are allowed to be re-screened, but enrollment will still require re-confirmation of inclusion criteria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy female Volunteers
Enrollment: 18000 (Actual)
Dates: Start 2023-08-13 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Combined Incidence of HPV Type 16/18-related CIN2/3, AIS, Invasive cervical cancer, VIN2/3, VaIN2/3, AIN1/2/3, vulvar, vaginal and anal cancer | 1 month after 3 doses of vaccine
  The endpoint is defined to have occurred: (a) a HPV Pathology Panel consensus diagnosis from the results of cervical biopsy: Cervical Intraepithelial Neoplasia (CIN, including grade 2 or 3), Adenocarcinoma in Situ (AIS), Invasive cervical cancer, Vulvar Intraepithelial Neoplasia (VIN, including grade 2 or 3), Vaginal Intraepithelial Neoplasia (VaIN, including grade 2 or 3), Anal intraepithelial neoplasia (AIN, including grade 1, 2, or 3), vulvar, vaginal and anal cancer; AND (b) detection of at least 1 of Human Papillomavirus (HPV) types 16/18 by Polymerase Chain Reaction (PCR) assay for virus subtype.
Combined Incidence of HPV Type 31/33/45/52/58-related CIN2/3, AIS, Invasive cervical cancer, VIN2/3, VaIN2/3, AIN1/2/3, vulvar, vaginal and anal cancer | 1 month after 3 doses of vaccine
  The endpoint is defined to have occurred: (a) a HPV Pathology Panel consensus diagnosis from the results of cervical biopsy: Cervical Intraepithelial Neoplasia (CIN, including grade 2 or 3), Adenocarcinoma in Situ (AIS), Invasive cervical cancer, Vulvar Intraepithelial Neoplasia (VIN, including grade 2 or 3), Vaginal Intraepithelial Neoplasia (VaIN, including grade 2 or 3), Anal intraepithelial neoplasia (AIN, including grade 1, 2, or 3), vulvar, vaginal and anal cancer; AND (b) detection of at least 1 of Human Papillomavirus (HPV) types 31/33/45/52/58 by Polymerase Chain Reaction (PCR) assay for virus subtype.
Combined Incidence of HPV Type 35/39/51/56/59-related CIN2/3, AIS, Invasive cervical cancer, VIN2/3, VaIN2/3, AIN1/2/3, vulvar, vaginal and anal cancer | 1 month after 3 doses of vaccine
  The endpoint is defined to have occurred: (a) a HPV Pathology Panel consensus diagnosis from the results of cervical biopsy: Cervical Intraepithelial Neoplasia (CIN, including grade 2 or 3), Adenocarcinoma in Situ (AIS), Invasive cervical cancer, Vulvar Intraepithelial Neoplasia (VIN, including grade 2 or 3), Vaginal Intraepithelial Neoplasia (VaIN, including grade 2 or 3), Anal intraepithelial neoplasia (AIN, including grade 1, 2, or 3), vulvar, vaginal and anal cancer; AND (b) detection of at least 1 of Human Papillomavirus (HPV) types 35/39/51/56/59 by Polymerase Chain Reaction (PCR) assay for virus subtype.

SECONDARY OUTCOMES:
Incidence of 6-month Persistent Infection associated with HPV types 16/18 | 1 month after 3 doses of vaccine
  The endpoint of a 6-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 2 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 6 months.
Incidence of 12-month Persistent Infection associated with HPV types 16/18 | 1 month after 3 doses of vaccine
  The endpoint of a 12-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 3 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 12 months.
Incidence of 6-month Persistent Infection associated with HPV types 31/33/45/52/58 | 1 month after 3 doses of vaccine
  The endpoint of a 6-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 2 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 6 months.
Incidence of 12-month Persistent Infection associated with HPV types 31/33/45/52/58 | 1 month after 3 doses of vaccine
  The endpoint of a 12-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 3 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 12 months.
Incidence of 6-month Persistent Infection associated with HPV types 35/39/51/56/59 | 1 month after 3 doses of vaccine
  The endpoint of a 6-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 2 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 6 months.
Incidence of 12-month Persistent Infection associated with HPV types 35/39/51/56/59 | 1 month after 3 doses of vaccine
  The endpoint of a 12-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 3 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 12 months.
Incidence of 6-month Persistent Infection associated with HPV types 6/11 | 1 month after 3 doses of vaccine
  The endpoint of a 6-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 2 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 6 months.
Incidence of 12-month Persistent Infection associated with HPV types 6/11 | 1 month after 3 doses of vaccine
  The endpoint of a 12-month Persistent Infection was defined to a subject was positive for the same HPV type by the HPV PCR assay to at least 1 common gene in 3 or more consecutive cervicovaginal/external genital swab, biopsy, or definitive therapy samples obtained for over a period of at least 12 months.
Incidence of histopathologically confirmed genital warts related to HPV types 6, 11 | 1 month after 3 doses of vaccine
  Genital warts were diagnosed by the HPV Vaccine program pathology panel from the results of cervical biopsy.
  HPV types 6/11 DNA was detected by PCR assay.
Incidence of histopathologically confirmed cervical, and/or anal, and/or vulvar, and/or vaginal lesions cases associated with HPV types 6/11/16/18 infection detected in the cervical cytology specimen | 1 month after 3 doses of vaccine
  HPV types 6/11/16/18 DNA was detected by PCR assay. Cervical, anal, vulvar, and vaginal lesions were diagnosed by the HPV vaccine program pathology panel from the results of cervical biopsy.
Incidence of histopathologically confirmed cervical, and/or anal, and/or vulvar, and/or vaginal lesions cases associated with HPV types 31/33/45/52/58 infection detected in the cervical cytology specimen | 1 month after 3 doses of vaccine
  HPV types 31/33/45/52/58 DNA was detected by PCR assay. Cervical, anal, vulvar, and vaginal lesions were diagnosed by the HPV vaccine program pathology panel from the results of cervical biopsy.
Incidence of histopathologically confirmed cervical, and/or anal, and/or vulvar, and/or vaginal lesions cases associated with HPV types 35/39/51/56/59 infection detected in the cervical cytology specimen | 1 month after 3 doses of vaccine
  HPV types 35/39/51/56/59 DNA was detected by PCR assay. Cervical, anal, vulvar, and vaginal lesions were diagnosed by the HPV vaccine program pathology panel from the results of cervical biopsy.
Incidence of histopathologically confirmed cervical, and/or anal, and/or vulvar, and/or vaginal lesions cases associated with HPV types 6/11/16/18/31/33/45/52/58 infection detected in the cervical cytology specimen | 1 month after 3 doses of vaccine
  HPV types 6/11/16/18/31/33/45/52/58 DNA was detected by PCR assay. Cervical, anal, vulvar, and vaginal lesions were diagnosed by the HPV vaccine program pathology panel from the results of cervical biopsy.
Incidence of histopathologically confirmed cervical, and/or anal, and/or vulvar, and/or vaginal lesions cases associated with HPV types 6/11/16/18/31/33/45/52/58/35/39/51/56/59 infection detected in the cervical cytology specimen | 1 month after 3 doses of vaccine
  HPV types 6/11/16/18/31/33/45/52/58/35/39/51/56/59 DNA was detected by PCR assay.
  Cervical, anal, vulvar, and vaginal lesions were diagnosed by the HPV vaccine program pathology panel from the results of cervical biopsy.
GMC of total anti-HPV6/11/16/18/31/33/45/52/58/35/39/51/56/59 type-associated specific IgG antibodies assessed by cLIA | At least 1 month after 3 doses of immunization
  GMCs was as geometric mean concertration of HPV Immunoglobulin G (IgG) antibodies and was measured using a Competitive Luminex Immunoassay (cLIA).
Positive conversion rate of total anti-HPV6/11/16/18/31/33/45/52/58/35/39/51/56/59 type-associated specific IgG antibodies assessed by cLIA | At least 1 month after 3 doses of immunization
  Positive conversion rate of total HPV6/11/16/18/31/33/45/52/58/35/39/51/56/59 type-associated specific IgG antibodies using cLIA.
GMT of HPV6/11/16/18/31/33/45/52/58/35/39/51/56/59 type-associated neutralizing antibodies. | At least 1 month after 3 doses of immunization
  GMTs was defined as geometric mean titers of HPV types 6/11/16/18/31/33/45/52/58/35/39/51/56/59 determined by pseudovirus-based neutralization assay.
AEs Incidence | During the entire study period (From Month 0 up to Month 60)
  Adverse Events (AEs) was considered to be all adverse medical events occurring after the subject is immunized with the experimental vaccine, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but are not necessarily causal to the experimental vaccine immunization relationship
SAEs Incidence | During the entire study period (From Month 0 up to Month 60)
  Serious Adverse Events (SAEs) was refered to adverse medical events, e.g., death, life-threatening, permanent or serious disability or loss of function, hospitalization or prolonged hospitalization of the subject, or congenital abnormality or birth defect after receiving the investigational vaccine. In addition, other important medical events should also be considered for SAE accelerated reporting
Pregnancy outcomes in pregnant subjects( pregnancy event report form) | During the entire study period (From Month 0 up to Month 60)
  Previous pregnancy, current pregnancy mode, neonatal information.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Mo, Principal Investigator — Guangxi Center for Disease Control and Prevention; Yan Zheng, Principal Investigator — Yunnan Center for Disease Control and Prevention; Guohua Li, Principal Investigator — Centers for Disease Control and Prevention, China; Ting Huang, Principal Investigator — Sichuan Center for Disease Control and Prevention; Zhiqaing Xie, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (5):
- China (5):
  - Guangxi Center for Disease Control and Prevention, Nanning, Guangxi
  - Henan Center for Disease Control and Prevention, Zhengzhou, Henan
  - Shanxi Center for Disease Control and Prevention, Taiyuan, Shanxi
  - Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan
  - Yunan Center for Disease Control and Prevention, Kunming, Yunan

IPD SHARING:
Plan to Share IPD: No